CLINICAL TRIAL: NCT01961622
Title: An Open-label, Multi-centre, Randomised, Two-period, Crossover Study to Assess the Efficacy, Safety and Utility of 12 Week Day and Night Automated Closed-loop Glucose Control Under Free Living Conditions Compared to Conventional Insulin Pump Therapy Combined With Continuous Glucose Monitoring in Adults With Type 1 Diabetes With Sub-optimal Glucose Control
Brief Title: Closing the Loop in Adults With Sub-optimally Controlled Type 1 Diabetes Under Free Living Conditions
Acronym: AP@home04
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry); Medical University of Graz (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Director of Research, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AP@home04
Record Dates: First submitted 2013-08-30; First posted 2013-10-11 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Closed loop insulin delivery; Continuous subcutaneous glucose monitoring; Continuous subcutaneous insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Florence D2A Closed Loop Glucose control (Experimental): Subjects glucose levels are controlled by Florence D2A or similar closed loop insulin delivery system
  Interventions: Device: Florence D2A or similar closed loop glucose control system
- CSII with real-time CGM (Active Comparator): Subject glucose level controlled by usual insulin pump therapy in conjunction with real time continuous glucose monitoring (FreeStyle Navigator CGM)
  Interventions: Device: CSII with real-time CGM

INTERVENTIONS:
Device: Florence D2A or similar closed loop glucose control system — Subject's glucose level will be controlled by the Florence D2A or similar automated closed loop glucose control system. The system comprises of FreeStyle Navigator 2 ® Continuous Glucose Monitoring (CGM) System (Abbott Diabetes Care, Alameda, CA, USA), Dana R Diabecare subcutaneous insulin infusion pump (Sooil Corp. Seoul, South Korea)or similar insulin pump, and MPC-based glucose control algorithm running on a smartphone
  Arms: Florence D2A Closed Loop Glucose control
Device: CSII with real-time CGM — Subject glucose level controlled by usual insulin pump therapy in conjunction with real time continuous glucose monitoring (CGM)
  Arms: CSII with real-time CGM

SUMMARY:
The main objective of this study is to determine whether day and night closed-loop insulin delivery for 12 weeks under free living conditions is superior to addition of real-time continuous glucose monitoring in adults with type 1 diabetes and sub-optimal glucose control on insulin pump therapy.

This is an open-label, multi centre, randomised, crossover design study, involving a 6 to 8 week run-in period, during which glucose control will be optimised by a professional pump educator, followed by two 3 months study periods during which glucose levels will be controlled either by an automated closed-loop system or by subjects usual insulin pump therapy augmented with real-time continuous glucose monitoring in random order. A total of up to 42 adults (aiming for 30 completed subjects) aged 18 years and older with T1D on insulin pump therapy will be recruited through diabetes clinics and other established methods in participating centres. Subjects who drop out of the study within the first 6 weeks of the first intervention arm will be replaced.

Subjects will receive appropriate training in the safe use of closed-loop insulin delivery system. Subjects will have regular contact with the study team during the home study phase including 24/7 telephone support. Subjects will be discouraged from international travel during the first two weeks of closed-loop use.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L as recorded by CGM (adjusted for potential over-estimation) during home stay. Secondary outcomes are the HbA1c, time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has type 1 diabetes as defined by WHO
2. The subject is 18 years of age or older
3. The subject will have been on an insulin pump for at least 6 months with good knowledge of insulin self-adjustment including carbohydrate counting
4. The subject is treated with one of the rapid acting insulin analogues (Insulin Aspart, Insulin Lispro or Insulin Glulisine)
5. HbA1c ≥7.5% (58mmol/mmol) and ≤ 10% (86 mmol/mmol) based on analysis from central laboratory or equivalent
6. The subject is willing to perform regular finger-prick blood glucose monitoring, with at least 6 measurements per day
7. The subject is willing to wear closed-loop system at home and at work place
8. The subject is willing to follow study specific instructions
9. The subject is willing to upload pump and CGM data at regular intervals
10. Female subjects of child bearing age should be on effective contraception and must have a negative urine-HCG pregnancy test at screening. In addition in Germany, women of childbearing potential must use a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e. less than 1% per year) and must use two independent methods of contraception, e.g. diaphragm and spermicide-coated condom.

Exclusion Criteria:

1. Non-type 1 diabetes mellitus
2. Any other physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results
3. Current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticosteroids, as judged by the investigator
4. Known or suspected allergy against insulin
5. Subjects with clinically significant nephropathy, neuropathy or proliferative retinopathy as judged by the investigator
6. Significantly reduced hypoglycaemia awareness as judged by the investigator
7. More than one episode of severe hypoglycaemia as defined by American Diabetes Association (31) in preceding 6 months (Severe hypoglycaemia is defined as an event requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions).
8. Random C-peptide > 100pmol/l with concomitant plasma glucose >4 mM(72 mg/dl)
9. Total daily insulin dose > 2 IU/kg/day
10. Subject is pregnant or breast feeding or planning pregnancy in near future (within next 3 months)
11. Severe visual impairment
12. Severe hearing impairment
13. Subjects using implanted internal pacemaker
14. Lack of reliable telephone facility for contact
15. Subject not proficient in English (UK) or German (Germany and Austria)
16. Subjects who are living alone

Additional exclusion criteria specific for Austria and Germany

1. Positive results on urine drug screen (amphetamines/metamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
2. Positive alcohol breath test.

Additional exclusion criteria specific for Germany only

1. Positive reaction to any of the following tests: hepatitis B surface (HBs) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus (HIV) 1 antibodies, anti-HIV2 antibodies.
2. Significantly reduced hypoglycaemia awareness withGold score ≥ 4 according to Geddes J et al, Diabetes Care 2007
3. Serious macro- and microangiopathy
4. Serious anomalies of the skin
5. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) located at places of the body, which potentially are possible to be used for localisation of the glucose sensor)
6. Renal insufficiency
7. Epilepsy
8. Eating disorders (like bulimia or anorexia nervosa)
9. Disorders of the lipid metabolism
10. Blood transfusion requiring patients
11. Psychiatric diseases and related conditions
12. Patients with frequent catheter abscesses having occurred in connection with the pump therapy
13. Patients with medically documented allergy towards the adhesive (glue) of plasters
14. Abnormal blood values for:

    * the creatinine clearance,
    * erythropoietin,
    * TSH.
15. Patients with the following concomitant medications or misuse of substances:

    * steroids,
    * anticoagulant therapies.
16. Patients with a planned intervention under general anaesthesia.
17. Patients who do shift work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time spent in the target glucose range from 3.9 to 10.0 mmol/l based on subcutaneous glucose monitoring | 90 days
  Time spent in the target glucose range from 3.9 to 10.0 mmol/l based on subcutaneous glucose monitoring (CGM) during the 90 days of home stay. Intention to treat basis.

SECONDARY OUTCOMES:
HbA1c | 90 days
  Measure of average glycaemic control during study period
Insulin dose | 90 days
  Total, basal and bolus insulin dose during 90 days of home periods
Adverse Events | 10 months
  Safety evaluation will comprise the number of episodes of hypoglycaemia, significant ketonemia (> 3.0mmol/l)as well as nature and severity of any other adverse events
Utility Evaluation | 90 days
  Utility evaluation is the frequency and duration of use of the closed-loop system at home and time between failures of closed-loop system components.
Continuous subcutaneous glucose monitoring (CGM) based outcome | 90 days
  Time spent above and below the target glucose 3.9 to 10.0 mmol/l, during the 90 days of home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 90 days
  Average,standard deviation and coefficient of variation of glucose levels during 90 days of home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 90 days
  The time with glucose levels < 3.5 mmol/l and <2.8 mmol/l during 90 days of home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 90 days
  The time with glucose levels in the significant hyperglycaemia,(glucose levels > 16.7 mmol/l during 90 days of home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 90 days
  Low Blood Glucose Index during 90 days of home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 90 days
  Duration of periods when sensor glucose values was below 3.5mmol/l for at least 20 minutes
Continuous subcutaneous glucose monitoring (CGM) based outcome | 90 days
  The "Area Under the Curve" below 3.5 mmol/l during 90 days home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 90 days
  Between 24 hour period variability: Coefficient of variation of CGM glucose between 24 hour periods (midnight to midnight)
Continuous subcutaneous glucose monitoring (CGM) based outcome | 90 days
  Glucose concentration in the target range (3.9-10.0mmol/L), and above and below target range based on adjusted CGM. Adjustment described in Hovorka R et. al.; Diabetes Technol Ther 14:1-9, 2012
Continuous subcutaneous glucose monitoring (CGM) based outcome during overnight period between 23:00 and 08:00 | 90 days
  Time spent with CGM glucose concentration in the target range (3.9-8.0mmol/L), Mean CGM glucose levels, The AUC below 3.5mmol/l, CV of CGM glucose levels, Coefficient of variation of CGM glucose between nights and Total insulin dose during overnight period between 23:00 and 08:00
Continuous subcutaneous glucose monitoring (CGM) based outcome during day period between 08:00 to 23:00 | 90 days
  Time spent with CGM glucose concentration in the target range (3.9-10.0mmol/L), Mean CGM glucose levels, The AUC below 3.5mmol/l, CV of CGM glucose levels, Coefficient of variation of CGM glucose between days and Total insulin dose during day period between 08:00 to 23:00

OTHER OUTCOMES:
Accuracy of CGM | 90 days
  CGM accuracy during 3 months home period; Capillary glucose vs. CGM will be evaluated using standard measures of numerical and clinical accuracy including absolute relative deviation and error grid analysis
Per Protocol Analysis | 90 days
  Per protocol analysis will be conducted to explore the relationship between usage of study treatments and study outcomes.
Effect of study intervention based on pre-study glycaemic control | 90 days
  Following outcomes will be calculated separately for participants with baseline HbA1c <8.5% vs. ≥ 8.5%
  Time spent with CGM glucose concentration in the target range (3.9-10.0mmol/L), Time spent with CGM glucose levels in hypoglycaemic range (< 3.9 mmol/L), Time spent with CGM glucose levels in hyperglycaemic range (> 10.0 mmol/L), Mean CGM glucose levels and the AUC below 3.5mmol/l based on continuous subcutaneous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Principal Investigator — University of Cambridge
Locations (3):
- Medical University of Graz, Graz, Austria
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany
- University of Cambridge, Cambridge, United Kingdom

REFERENCES:
- [Background] Hovorka R, Allen JM, Elleri D, Chassin LJ, Harris J, Xing D, Kollman C, Hovorka T, Larsen AM, Nodale M, De Palma A, Wilinska ME, Acerini CL, Dunger DB. Manual closed-loop insulin delivery in children and adolescents with type 1 diabetes: a phase 2 randomised crossover trial. Lancet. 2010 Feb 27;375(9716):743-51. doi: 10.1016/S0140-6736(09)61998-X. Epub 2010 Feb 4. PMID 20138357
- [Background] Hovorka R, Kumareswaran K, Harris J, Allen JM, Elleri D, Xing D, Kollman C, Nodale M, Murphy HR, Dunger DB, Amiel SA, Heller SR, Wilinska ME, Evans ML. Overnight closed loop insulin delivery (artificial pancreas) in adults with type 1 diabetes: crossover randomised controlled studies. BMJ. 2011 Apr 13;342:d1855. doi: 10.1136/bmj.d1855. PMID 21493665
- [Background] Hovorka R. Closed-loop insulin delivery: from bench to clinical practice. Nat Rev Endocrinol. 2011 Feb 22;7(7):385-95. doi: 10.1038/nrendo.2011.32. PMID 21343892
- [Derived] Thabit H, Tauschmann M, Allen JM, Leelarathna L, Hartnell S, Wilinska ME, Acerini CL, Dellweg S, Benesch C, Heinemann L, Mader JK, Holzer M, Kojzar H, Exall J, Yong J, Pichierri J, Barnard KD, Kollman C, Cheng P, Hindmarsh PC, Campbell FM, Arnolds S, Pieber TR, Evans ML, Dunger DB, Hovorka R. Home Use of an Artificial Beta Cell in Type 1 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2129-2140. doi: 10.1056/NEJMoa1509351. Epub 2015 Sep 17. PMID 26379095
- [Derived] Leelarathna L, Dellweg S, Mader JK, Barnard K, Benesch C, Ellmerer M, Heinemann L, Kojzar H, Thabit H, Wilinska ME, Wysocki T, Pieber TR, Arnolds S, Evans ML, Hovorka R; AP@home consortium. Assessing the effectiveness of 3 months day and night home closed-loop insulin delivery in adults with suboptimally controlled type 1 diabetes: a randomised crossover study protocol. BMJ Open. 2014 Sep 3;4(9):e006075. doi: 10.1136/bmjopen-2014-006075. PMID 25186158